CLINICAL TRIAL: NCT02033811
Title: MitraClip® Registry - an Observational Study of Percutaneous Mitral Valve Repair Using the MitraClip® System
Brief Title: MitraClip® Registry
Status: Recruiting | Type: Observational
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Director Division of Cardiology, Pulmonary Disease and Vascular Medicine, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: MitraClip® Registry
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Mitral Regurgitation
Keywords: mitral regurgitation; MitraClip system; percutaneous mitral valve repair
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Percutaneous mitral valve repair with the MitraClip® system has emerged as a therapeutic alternative to surgical valve repair (PMVR) in high risk patients.

The aim of this registry is to collect prospectively and systematically clinical research data from patients undergoing PMVR with the MitraClip® system. This registry is an open-end observational study to assess the characteristics and outcomes patients with severe mitral regurgitation undergoing PMVR.

ELIGIBILITY:
Inclusion Criteria:

* severe mitral regurgitation
* percutaneous mitral valve repair (PMVR) with the MitraClip® system

Exclusion Criteria:

* < 18 years
* Patients considered by the heart team to be unlikely to receive meaningful or durable clinical benefit from the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing percutaneous mitral valve repair (PMVR) with the MitraClip® system
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Major cardiac adverse events | 30 days
  increase in the 30-day risk of adverse events among patients receiving PMVR

SECONDARY OUTCOMES:
Mortality | 1 year
  Proportion of patients who are alive at 1 year after receiving

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, MD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine; Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Heinrich Heine University Div. of Cardiology, Pulmonary Disease and Vasculae Medicine, Düsseldorf, Germany

REFERENCES:
- [Derived] Herbrand T, Eschenhagen S, Zeus T, Kehmeier E, Hellhammer K, Veulemans V, Kelm M, Balzer J. Acute reverse annular remodeling during MitraClip(R) therapy predicts improved clinical outcome in heart failure patients: a 3D echocardiography study. Eur J Med Res. 2017 Sep 20;22(1):33. doi: 10.1186/s40001-017-0273-x. PMID 28931437
- [Derived] Rammos C, Zeus T, Balzer J, Veulemans V, Hellhammer K, Niebel S, Kelm M, Rassaf T. Left Atrial and Left Ventricular Function and Remodeling Following Percutaneous Mitral Valve Repair. J Heart Valve Dis. 2016 May;25(3):309-319. PMID 27989041
- [Derived] Hellhammer K, Zeus T, Balzer J, van Hall S, Rammos C, Wagstaff R, Kelm M, Rassaf T. Safety and efficacy of percutaneous mitral valve repair using the MitraClip(R) system in patients with diabetes mellitus. PLoS One. 2014 Nov 6;9(11):e111178. doi: 10.1371/journal.pone.0111178. eCollection 2014. PMID 25375257
- See also: Related Info — http://www.uniklinik-duesseldorf.de/kardiologie